CLINICAL TRIAL: NCT06829043
Title: Utilizzo Della 18F-FDG PET/TC Per Stratificare Il Rischio Di Malignità Dei Noduli Tiroidei a Citologia Indeterminata (TIR3A E TIR3B)
Brief Title: 18F-FDG PET/TC in TIR3A E TIR3B
Acronym: PET-TIR3-2021
Status: Enrolling by invitation | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: 50/2022/Oss/AOUBo; 50/2022/Oss/AOUBo (Registry Identifier: AOSP Bologna)
Record Dates: First submitted 2025-02-11; First posted 2025-02-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2024-12

CONDITIONS: PET / CT; FDG PET/CT; Cytology; Thyroid Nodules
Keywords: PET/TC; cytology; 18F-FDG; thyroid nodules
MeSH Terms: conditions — Thyroid Nodule

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- TIR3 group: The study is addressed to all patients belonging to the U.O. of Nuclear Medicine of the IRCCS AOU of Bologna for execution of needle aspirate on thyroid nodules with undetermined cytology (TIR3A, TIR3B) and candidates for surgery from 1 February 2022 to 1 February 2027. These patients will be referred to 18F-FDG PET/CT survey at our Center. If the patient has already performed the 18F-FDG PET/CT survey at our Center (within 4 months of performing the needle aspiration), with guidelines, this survey will be included without repetition.
  Interventions: Other: clinical practice drug treatment

INTERVENTIONS:
Other: clinical practice drug treatment — The study is observational, non-interventional and involves the review of the investigation18F-FDGPET/TC (performed according to the EANM guidelines) by two experts from the Nuclear Medicine Department.

SUMMARY:
The primary objective of this study is to evaluate the diagnostic performance of 18F-FDG PET/CT performed by normal care pathway in the identification of malignancy of undetermined resulting thyroid lesions at cytology (TIR3A and TIR3B) comparing the 18F-FDG PET/CT result with histological data.

The secondary objective is to identify possible PET/ultrasound/genetic/radiomics variables that can more accurately define the potential malignancy of undetermined nodules and create a predictive model of malignity fed by standard parameters (derived from the normal care path).

The identification of the prognostic value of 18F-FDG PET/CT in such patients setting could, in fact, make the PET useful in the future in the selection of patients for surgery/ follow-up.

DETAILED DESCRIPTION:
To better stratify the malignancy risk of the resulting undetermined cytological lesions (TIR3A and TIR3B), it is proposed to perform an 18F-FDG PET/TC survey in these patients by which semiquantitative parameters are derived (SUVmax, SUVmean, SUVpeak, MTV, TLG) and perform radiomatic analysis. In the case where the above mentioned PET/CT survey has been recently performed, the survey will not be repeated but the images will be reviewed with visual and semi-quantitative analysis. The results will be compared with those derived from ultrasound and genetic analysis (currently proposed in cases of TIR3A), with the subsequent histological examination derived from surgery (currently indicated by the normal care path in TIR3B cases and in case of reconfirmation of TIR3A cytology to a second needle aspiration on the nodule). It is expected that an algorithm with multiple parameters combined can be created to correctly point towards surgery or a conservative attitude of follow up.

ELIGIBILITY:
Inclusion Criteria:

* Patients with undetermined cytology (TIR3B and TIR3A candidates for surgery) and 18F-FDG PET/CT;
* Obtaining informed consent for data collection and processing.
* Patient aged 18 years

Exclusion Criteria:

- Pregnant/breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study is addressed to all patients belonging to the U.O. of Nuclear Medicine of the IRCCS AOU of Bologna for execution of needle aspirate on thyroid nodules with undetermined cytology (TIR3A, TIR3B) and candidates for surgery from 1 February 2022 to 1 February 2027. These patients will be referred to 18F-FDG PET/CT survey at our Center. If the patient has already performed the 18F-FDG PET/CT survey at our Center (within 4 months of performing the needle aspiration), with guidelines, this survey will be included without repetition.
  The expected duration of the scientific study (patient enrollment, data analysis, preparation of an article) is 6 years.
Sampling Method: Probability Sample
Enrollment: 216 (Estimated)
Dates: Start 2022-03-22 (Actual); Primary Completion 2024-12-12 (Actual); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
diagnostic performance | 6 years
  the diagnostic capacity of 18F-FDG PET/CT evaluated by calculating the percentages of true positives, false positives, true negatives and false negatives through comparison between the histological data (positivity or negativity for neoplasm) with the 18F-FDG PET/CT (positivity or negativity to PET/CT images).

CONTACTS AND LOCATIONS:
Locations (1):
- Nuclear medicine, IRCCS, Azienda Ospedalierio-Universitaria di Bologna, Bologna, Italy, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kresnik E, Gallowitsch HJ, Mikosch P, Stettner H, Igerc I, Gomez I, Kumnig G, Lind P. Fluorine-18-fluorodeoxyglucose positron emission tomography in the preoperative assessment of thyroid nodules in an endemic goiter area. Surgery. 2003 Mar;133(3):294-9. doi: 10.1067/msy.2003.71. PMID 12660642
- [Background] Abooshahab R, Gholami M, Sanoie M, Azizi F, Hedayati M. Advances in metabolomics of thyroid cancer diagnosis and metabolic regulation. Endocrine. 2019 Jul;65(1):1-14. doi: 10.1007/s12020-019-01904-1. Epub 2019 Apr 1. PMID 30937722